CLINICAL TRIAL: NCT04252898
Title: Impact of a Front-of-pack Nutrition Labelling on the Nutritional Quality of Purchases of Customers in Contract Catering - a Controlled Trial
Brief Title: Impact of a Front-of-pack Nutrition Labelling on Food Purchases in Contract Catering
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Paris 13 (Other)
Collaborators: ELIOR GESTION (Unknown)
Responsible Party: Principal Investigator, Mathilde Touvier, Professor, University of Paris 13
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: ELIOR
Record Dates: First submitted 2020-01-24; First posted 2020-02-05 (Actual); Last update posted 2021-08-06 (Actual); Status verified 2021-08

CONDITIONS: Food Labeling
Keywords: Food labeling; nutritional quality; food purchases

STUDY DESIGN:
Intervention Model Description: The trial will include four sites (two pairs, with an intervention site and a control site) and two phases.
  For each pair of sites:
  * site n°1: one control phase with no intervention followed by an interventional phase with the Nutri-Score applied on products
  * site n°2: control phases only, without the Nutri-Score applied during any of the two phases
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention arm (Experimental): In this arm (site n°1), participants will purchase their products in the restaurant first in a control phase and then in an interventional phase with the Nutri-Score affixed on food products.
  Interventions: Behavioral: Front-of-pack nutrition label Nutri-Score
- Control arm (No Intervention): In this arm (site n°2), participants will purchase their products in the restaurant during the whole study without any label affixed on food products.

INTERVENTIONS:
Behavioral: Front-of-pack nutrition label Nutri-Score — The intervention consists of displaying the Nutri-Score on dishes and pre-packed foods.
  Arms: Intervention arm

SUMMARY:
This controlled trial investigates the impact of the implementation of a front-of-pack nutrition label, namely Nutri-Score, on foods and beverages sold in a contract catering in France on the nutritional quality of purchases.

DETAILED DESCRIPTION:
The introduction of front-of-pack nutrition labelling is thought to help consumers making healthier food choices at the point-of-purchase. In 2017, the French government has selected the Nutri-Score as single front-of-pack nutrition label to be applied on food products sold in French supermarkets, on a voluntary basis.

Some studies have found that the Nutri-Score would help consumers making healthier choices. Nevertheless, its impact has been demonstrated in experimental supermarkets and its implementation only concerns products sold in groceries and supermarkets, as it is stated in the official decree. The potential impact of the Nutri-Score in contract catering remains unknown, while this sector represents a growing share of out-of-home catering and that the promotion of the Nutri-Score in this sector is now part of the National Public Health Plan.

Thus, the objective of the present study is to investigate the impact of the implementation of the Nutri-Score in contract catering restaurants on the nutritional quality of food purchases. The trial will be conducted using a quasi experimental before/after design with a comparison group. Data on purchases will be collected regularly through receipts, and the nutritional quality of purchases will be evaluated over time on two pairs of sites. In each pair of sites, one site will receive an intervention (Nutri-Score) and one site will be a control site. Within each pair, the sites will be comparable in terms of food offer and consumers profile.

ELIGIBILITY:
Inclusion Criteria:

* all individuals purchasing in the contract catering restaurants will be included.

Exclusion Criteria:

* No

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 2082 (Actual)
Dates: Start 2019-12-16 (Actual); Primary Completion 2020-03-13 (Actual); Study Completion 2020-03-13 (Actual)

PRIMARY OUTCOMES:
Change in the overall nutritional quality of purchases over time | Through study completion, an average of 6 months
  Score using the Food Standards Agency nutrient profiling system modified by the HCSP, allocating points depending on the amounts in unfavourable elements (energy, saturates, sugars, sodium) and favorable elements (fibres, proteins and fruits, vegetables, nuts and oils (olive, colza, nuts))

SECONDARY OUTCOMES:
Change in energy content of purchases | Through study completion, an average of 6 months
  Energy content of the purchases in kcal / 100g
Change in Saturated fat content of purchases | Through study completion, an average of 6 months
  Saturated fat content of the purchases in g / 100g
Change in Sugar content of purchases | Through study completion, an average of 6 months
  Sugar content of the purchases in g / 100g
Change in Sodium content of purchases | Through study completion, an average of 6 months
  Sodium content of the purchases in mg / 100g
Change in Protein content of purchases | Through study completion, an average of 6 months
  Protein content of the purchases in g / 100g
Change in Fibre content of purchases | Through study completion, an average of 6 months
  Fibre content of the purchases in g / 100g
Change in Fruit, vegetable and nut content of purchases | Through study completion, an average of 6 months
  Fruit, vegetable and nut content of the purchases in % / 100g

CONTACTS AND LOCATIONS:
Locations (1):
- Equipe de Recherche en Epidémiologie Nutritionnelle, Bobigny, France